CLINICAL TRIAL: NCT03057808
Title: Gestational Weight Gain and Postpartum Weight Loss in Active Duty Women
Brief Title: Gestational Weight Gain and Postpartum Weight Loss in Active Duty Women (Moms Fit 2 Fight)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Tennessee (Other)
Collaborators: 59th Medical Wing (U.S. Federal Agency); San Antonio Military Medical Center (U.S. Federal Agency); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 16-04804-XP DOD; 1R01DK104872-01A1 (NIH)
Record Dates: First submitted 2017-01-03; First posted 2017-02-20 (Actual); Results first posted 2022-12-23 (Actual); Last update posted 2022-12-23 (Actual); Status verified 2022-07

CONDITIONS: Weight Gain; Weight Loss
Keywords: Pregnancy; Postpartum
MeSH Terms: conditions — Weight Gain; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Gestational weight gain intervention (GWG-only) (Experimental): The GWG intervention will begin upon randomization to the GWG-only or the GWG+PPWL arm, and continue until the birth of the participant's child.
  Interventions: Behavioral: Gestational weight gain intervention
- Postpartum weight loss intervention (PPWL-only) (Experimental): The PPWL intervention will begin at 6-weeks postpartum (when most women will be approved for weight loss and exercise by their obstetrician) for those participants randomized to the PPWL only or the GWG+PPWL arms, and will continue until 6-months postpartum.
  Interventions: Behavioral: Postpartum weight loss intervention
- Combined (Experimental): During the gestational phase participants will receive the same intervention as the GWG only group. During the postpartum phase participants will receive the the same intervention as the PPWL group.
  Interventions: Behavioral: Gestational weight gain intervention; Behavioral: Postpartum weight loss intervention

INTERVENTIONS:
Behavioral: Gestational weight gain intervention — This intervention will provide individual, telephone-based sessions (20-30 minutes each) by trained interventionists. The intervention will focus on self-monitoring, clear goals (i.e., GWG, caloric intake exercise), and problem solving.
  Other Names: GWG-only
  Arms: Combined; Gestational weight gain intervention (GWG-only)
Behavioral: Postpartum weight loss intervention — The PPWL intervention will provide individual, telephone-based sessions (20-30 minutes each) by trained interventionists. (The number of possible telephone sessions will depend on the level of support needed by each participant to meet her weight loss goals). The PPWL intervention will focus on self-monitoring; weight, dietary intake and exercise goals; and problem solving.
  Other Names: PPWL-only
  Arms: Combined; Postpartum weight loss intervention (PPWL-only)

SUMMARY:
The purpose of this study is to enroll approximately 450 subjects to see if a behavioral weight management program is successful in helping TRICARE beneficiaries who are pregnant or post-partum to manage their weight during and after their pregnancy.

DETAILED DESCRIPTION:
Investigators will randomize 450 consented participants to 1 of 3 interventions: a) a gestational weight gain intervention (GWG-only); b) a postpartum weight loss intervention (PPWL-only), or c) a combined gestational weight gain and postpartum weight loss intervention (GWG+PPWL) to determine the efficacy of the interventions on GWG as well as PPWL.

Procedures: Interested individuals will be directed to call the study telephone number to learn more and determine whether eligibility criteria is met. Individuals who meet the telephone screening eligibility criteria will be invited to schedule a Screening Visit, during which written informed consent will be obtained. At this visit, eligibility will be assessed and measures will be administrated. The potential participant will also be asked to complete a one-week dietary and exercise self-monitoring run-in and receive medical clearance from their obstetrician to participate. Should she continue to be interested, she will return for a Baseline Visit and will be randomized.

Randomized participants will have 5 in person scheduled visits after their Screening Visit and Baseline Visit to the Wilford Hall Ambulatory Surgical Center (WHASC) or San Antonio Military Medical Center (SAMMC) Obstetrics (OB) clinic. These visits will be scheduled at gestational week 32, 36, as well as at 6- weeks, 6-months, and 12- month postpartum. At these visits, physical measurements will be collected and participants will complete various questionnaires.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be active duty military, dependents or retired with TRICARE benefits
* Participants must be less than 12 weeks gestation upon recruitment (based on the date of their last menstrual period and then confirmed by their physician at their first prenatal visit, which typically occurs at 6-8 weeks gestation at WHASC and SAMMC)
* Participants also must be within the normal, overweight, or obese BMI ranges
* Are generally in good health
* Currently not smoking more than 5 cigarettes per day at the time of conception

Exclusion Criteria:

* Expecting multiple babies (e.g. twins)
* Diabetic
* Not interested in participating in a program for 21 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 430 (Actual)
Dates: Start 2017-02-06 (Actual); Primary Completion 2021-11-10 (Actual); Study Completion 2022-05-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Krukowski, PhD, Principal Investigator — University of Tennessee
Locations (2):
- United States (2):
  - San Antonio Military Medical Center Obstetrics Clinic (SAMMC), San Antonio, Texas
  - Wilford Hall Ambulatory Surgical Center, San Antonio, Texas

REFERENCES:
- [Derived] Solomon E, McPhail A, Bursac Z, Little MA, Talcott GW, Krukowski RA. Provider advice, pregnant persons' expectations, and actual gestational weight gain among United States military health care beneficiaries: a secondary analysis of a randomized controlled trial. BMC Pregnancy Childbirth. 2024 Nov 25;24(1):785. doi: 10.1186/s12884-024-06987-x. PMID 39587506
- [Derived] Perez-Munoz A, Hare ME, Andres A, Klesges RC, Wayne Talcott G, Little MA, Waters TM, Harvey JR, Bursac Z, Krukowski RA. A Postpartum Weight Loss-focused Stepped-care Intervention in a Military Population: A Randomized Controlled Trial. Ann Behav Med. 2023 Sep 13;57(10):836-845. doi: 10.1093/abm/kaad014. PMID 37061829
- [Derived] Pebley K, Farage G, Hare ME, Bursac Z, Andres A, Chowdhury SMR, Talcott GW, Krukowski RA. Changes in self-reported and accelerometer-measured physical activity among pregnant TRICARE Beneficiaries. BMC Public Health. 2022 Nov 7;22(1):2029. doi: 10.1186/s12889-022-14457-2. PMID 36336697
- [Derived] Estevez Burns R, Hare ME, Andres A, Klesges RC, Talcott GW, LeRoy K, Little MA, Hyrshko-Mullen A, Waters TM, Harvey JR, Bursac Z, Krukowski RA. An interim analysis of a gestational weight gain intervention in military personnel and other TRICARE beneficiaries. Obesity (Silver Spring). 2022 Oct;30(10):1951-1962. doi: 10.1002/oby.23523. Epub 2022 Aug 30. PMID 36041980

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Initially, participants were required to receive obstetric care at either San Antonio Military Medical Center or Wilford Hall Ambulatory Surgical Center. With the obstetric clinic closure at Wilford Hall Ambulatory Surgical Center in October 2019 and the coronavirus pandemic, recruitment was expanded to include obstetric clinics at Andrews and Wright Patterson Air Force Bases in July 2020. Interested individuals were recruited between February 2017 to October 2020.
Pre-assignment Details: Potentially eligible participants presented for a screening visit where full eligibility was assessed, informed consent was obtained, and study measures were collected. Participants were then asked to track their diet and exercise for one week and obtain their obstetrician's clearance for participation. Active duty personnel were also required to submit their fitness test scores for the year prior to study enrollment, to facilitate comparisons with their postpartum fitness test scores.
Period: Overall Study
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Started | 144 | 142 | 144
32-36 Weeks Gestation | 129 | 129 | 120
Completed | 132 | 121 | 127
Not Completed | 12 | 21 | 17

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined | Total
Number analyzed (Participants) | 144 | 142 | 144 | 430
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.9 (4.9) | 30.4 (4.8) | 30.6 (4.8) | 30.6 (4.9)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 144 | 142 | 144 | 430
  Male | 0 | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 22 | 21 | 29 | 72
  Not Hispanic or Latino | 122 | 121 | 115 | 358
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 2 | 2
  Asian | 2 | 5 | 6 | 13
  Native Hawaiian or Other Pacific Islander | 2 | 0 | 3 | 5
  Black or African American | 20 | 22 | 22 | 64
  White | 101 | 99 | 92 | 292
  More than one race | 5 | 3 | 13 | 21
  Unknown or Not Reported | 14 | 13 | 6 | 33
Region of Enrollment [Number; unit: participants]
  United States | 144 | 142 | 144 | 430
Body mass index [Mean (Standard Deviation); unit: Kg/m^2] | 27.6 (5.3) | 27.7 (5.5) | 27.6 (5.0) | 27.6 (5.2)
Gestational week at screening [Mean (Standard Deviation); unit: weeks] | 11.8 (1.1) | 11.6 (1.2) | 11.8 (1.0) | 11.7 (1.1)
Active duty [Count of Participants; unit: Participants] | 70 | 64 | 70 | 204
Previous live birth [Count of Participants; unit: Participants] | 80 | 80 | 80 | 240

OUTCOME MEASURES:

1. Primary Outcome: Changes in the Mother's Body Weight Pre and Post Pregnancy
Description: At all measurement visits, weight will be recorded in kilograms. Weight will be measured on a calibrated digital scale in duplicate, with the participant wearing light clothing and no shoes. While Investigators obtain the mother's weight at baseline, there will also be a self reported pregravid weight (before the last menstrual period).
Time Frame: Baseline to 6 months postpartum
Population: Those who completed the 6 month postpartum visit
Measure: Mean (Standard Deviation); unit: kilograms
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Number analyzed (Participants) | 132 | 121 | 127
kilograms | 2.39 (5.36) | 1.25 (5.40) | 1.37 (5.76)

2. Secondary Outcome: Maternal and Fetal Conditions During Pregnancy
Description: Pregnancy-related medical outcomes will be obtained from the participant's medical record and will include: maternal (e.g., gestational diabetes, preeclampsia) and fetal conditions.
Time Frame: Baseline (13 weeks gestational to delivery)
Population: Those who delivered in military hospitals, with some missing data for some of the variables. The two conditions that received the same intervention during the gestational period (GWG-only, Combined) were combined for analyses and compared to the PPWL-only condition.
Measure: Count of Participants; unit: Participants
Groups:
- Participants Who Received the Gestational Weight Gain Intervention (GWG-only, Combined): The GWG intervention will begin upon randomization to the GWG-only or the GWG+PPWL arm, and continue until the birth of the participant's child.
  Gestational weight gain intervention: This intervention will provide individual, telephone-based sessions (20-30 minutes each) by trained interventionists. The intervention will focus on self-monitoring, clear goals (i.e., GWG, caloric intake exercise), and problem solving.
- Comparison Condition (PPWL-only): Participants who did not receive the GWG intervention
Arm/Group | Participants Who Received the Gestational Weight Gain Intervention (GWG-only, Combined) | Comparison Condition (PPWL-only)
Number analyzed (Participants) | 233 | 115
Participants
  Preeclampsia | 22 | 13
  Pregancy inducaed hypertension | 35 | 26
  Gestational diabetes | 17 | 13
  Cesarean delivery (elective) | 36 | 18
  Cesarean delivery (emergency) | 39 | 14
  Preterm delivery (<37 weeks) | 14 | 7
  Small-for-gestational age (<10th percentile) | 15 | 7
  Large-for-gestational age (> 90th percentile) | 19 | 9
  Neonatal Intensive Care Unit admission) | 19 | 12

3. Secondary Outcome: Birth Weight of Infant
Description: Birth weight of the infant will be recorded in grams.
Time Frame: Delivery
Population: For participants who delivered at a military hospital. The two conditions that received the same intervention during the gestational period (GWG-only, Combined) were combined for analyses and compared to the PPWL-only condition.
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | Participants Who Received the Gestational Weight Gain Intervention (GWG-only, Combined) | Comparison Condition (PPWL-only)
Number analyzed (Participants) | 225 | 106
grams | 3363.5 (529.1) | 3365.3 (545.8)

4. Secondary Outcome: Length of Infant
Description: Birth height of the infant will be recorded in centimeters.
Time Frame: Delivery
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: centimeters
Arm/Group | Participants Who Received the Gestational Weight Gain Intervention (GWG-only, Combined) | Comparison Condition (PPWL-only)
Number analyzed (Participants) | 209 | 100
centimeters | 51.3 (2.8) | 50.8 (4.0)

5. Secondary Outcome: Waist Circumference on Fitness Test Scores
Description: Waist circumference will be recorded in centimeters.
Time Frame: Baseline and 12 months postpartum
Population: Due to the coronavirus pandemic, military fitness tests were suspended for approximately 18 months, which did not allow for postpartum fitness tests to be conducted at the designated time.
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Number of Push Ups on Fitness Test Scores
Description: Number of push ups completed.
Time Frame: Baseline and 12 months postpartum
Population: Due to the COVID-19 pandemic, military fitness tests were suspended for approximately 18 months, which did not allow for postpartum fitness tests to be conducted at the designated time.
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Number analyzed (Participants) | 0 | 0 | 0

7. Secondary Outcome: Number of Sit Ups on Fitness Test Scores
Description: Number of sit ups completed.
Time Frame: Baseline and 12 months postpartum
Population: as for outcome 6
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Number analyzed (Participants) | 0 | 0 | 0

8. Secondary Outcome: 1.5 Mile Run on Fitness Test Scores
Description: The amount of time it took to complete 1.5 miles.
Time Frame: Baseline and 12 months postpartum
Population: as for outcome 6
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Number analyzed (Participants) | 0 | 0 | 0

9. Secondary Outcome: Moms Fit 2 Fight Program Evaluation Form
Description: Program satisfaction will be assessed using the Investigators program evaluation form to offer insight into program acceptability as well as barriers and facilitators to participation in each intervention arm. Participants will be given 10 statements to rate their experience using a 5 point scale.
Time Frame: 12 months postpartum
Population: Includes participants who completed the 12 month program satisfaction measure and did not indicate "don't know"
Measure: Count of Participants; unit: Participants
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
Number analyzed (Participants) | 111 | 103 | 109
Participants
  Found the program useful: number analyzed (Participants) | 109 | 101 | 109
  Found the program useful | 96 | 88 | 93
  Enjoyed the program: number analyzed (Participants) | 110 | 100 | 109
  Enjoyed the program | 95 | 87 | 96
  Would recommend the program: number analyzed (Participants) | 111 | 101 | 105
  Would recommend the program | 104 | 99 | 96
  Appropriate number of sessions: number analyzed (Participants) | 107 | 96 | 104
  Appropriate number of sessions | 90 | 85 | 93
  Appropriate length of sessions: number analyzed (Participants) | 107 | 97 | 106
  Appropriate length of sessions | 100 | 92 | 92
  Lesson materials were helpful: number analyzed (Participants) | 101 | 87 | 93
  Lesson materials were helpful | 82 | 75 | 71
  Diet/Exercise monitoring was helpful: number analyzed (Participants) | 107 | 96 | 106
  Diet/Exercise monitoring was helpful | 95 | 86 | 90
  Electronic scale was helpful: number analyzed (Participants) | 109 | 101 | 109
  Electronic scale was helpful | 104 | 98 | 109
  Meal replacements were helpful: number analyzed (Participants) | 39 | 35 | 41
  Meal replacements were helpful | 29 | 31 | 32
  Meal plans were helpful: number analyzed (Participants) | 42 | 38 | 38
  Meal plans were helpful | 31 | 29 | 27

ADVERSE EVENTS:
Time Frame: From study enrollment/consent to 12 months postpartum (approximately 20 months)
Description: At each data collection visit, the participants were asked if they experienced any changes in their health since the last visit
Arm/Group | Gestational Weight Gain Intervention (GWG-only) | Postpartum Weight Loss Intervention (PPWL-only) | Combined
All-Cause Mortality (participants affected / at risk) | 0/144 | 0/142 | 0/144
Serious Adverse Events (participants affected / at risk) | 23/144 | 13/142 | 22/144
Other Adverse Events (participants affected / at risk) | 30/144 | 38/142 | 46/144
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gestational Weight Gain Intervention (GWG-only) (N=144) | Postpartum Weight Loss Intervention (PPWL-only) (N=142) | Combined (N=144)
Appendectomy (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Tubal ligation (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 1 (1)
Preterm labor/delivery (Pregnancy, puerperium and perinatal conditions) | 7 (7) | 1 (1) | 3 (3)
Caesarean section (Reproductive system and breast disorders) | 6 (6) | 1 (1) | 3 (3)
Miscarriage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 4 (4) | 3 (3)
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 5 (5) | 3 (3) | 1 (1)
Kidney infection (Renal and urinary disorders) | 1 (1) | 1 (1) | 0 (0)
Syncope (General disorders) | 1 (1) | 0 (0) | 0 (0)
NICU admission (General disorders) | 1 (1) | 0 (0) | 1 (1)
Low white blood count (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Heart rate issues (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Gallbladder removal (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Hospitalization due to viral illness (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Kidney stones (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0)
Uterine bleeding (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 0 (0) | 0 (0)
Elevated blood pressure with amniotic fluid leak (General disorders) | 1 (1) | 0 (0) | 0 (0)
Chest pains, shortness of breath, syncope (General disorders) | 1 (1) | 0 (0) | 0 (0)
Placenta previa (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) | 0 (0)
Ruptured rectum (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Fetal Single Umbilical Artery (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0)
Epileptic event (Nervous system disorders) | 0 (0) | 1 (1) | 1 (1)
Retained placenta (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Car accident (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
Mastitis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Nausea and vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Gallbladder stone (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (1)
Dermoid cyst (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1)
Fetal termination due to anomalies (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 0 (0) | 1 (1)
Neonatal death (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Cellulitis infection (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Gestational Weight Gain Intervention (GWG-only) (N=144) | Postpartum Weight Loss Intervention (PPWL-only) (N=142) | Combined (N=144)
Common cold (Infections and infestations) | 9 (9) | 12 (12) | 20 (20)
Depressive symptoms (Psychiatric disorders) | 12 (12) | 14 (14) | 17 (17)
Gestational diabetes (Pregnancy, puerperium and perinatal conditions) | 11 (11) | 6 (6) | 13 (13)
Back pain (Musculoskeletal and connective tissue disorders) | 4 (4) | 3 (3) | 10 (10)
COVID-19 (Infections and infestations) | 2 (2) | 8 (8) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-01-03): https://cdn.clinicaltrials.gov/large-docs/08/NCT03057808/Prot_SAP_000.pdf